CLINICAL TRIAL: NCT07030647
Title: Efficacy of the Analgesic Effect of Local Anesthetic Injection on Postoperative Pain in Gynecological Laparoscopic Surgeries: A Randomized Controlled Trial
Brief Title: "Efficacy of Local Anesthetic for Postoperative Pain in Gynecologic Laparoscopy"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Usama Ahmed Elsaeed Salem, MD (Other)
Responsible Party: Sponsor-Investigator, Usama Ahmed Elsaeed Salem, MD, Usama Ahmed Elsaeed Salem, MD, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Cairo University., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-447-2024
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Gynecologic Laparoscopic Surgery; Postoperative Pain; Recovery Outcomes; Pain Management
Keywords: Gynecological laparoscopy, local anesthetic infiltration, postoperative pain, recovery, bupivacaine, port-site infiltration; Intraperitoneal local anesthetic
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Port Site Local Anesthetic Injection (Group A) (Experimental): Participants receive a local anesthetic injection at the trocar/port sites of laparoscopic gynecologic surgery.
  Interventions: Drug: Bupivacaine 0.25%
- Intraperitoneal Local Anesthetic Injection (Group B) (Experimental): Participants receive an intraperitoneal local anesthetic injection before removal of the laparoscopic instruments.
  Interventions: Drug: Bupivacaine 0.25%
- Control (Group C) (No Intervention): Participants receive no local anesthetic injection during surgery.

INTERVENTIONS:
Drug: Bupivacaine 0.25% — At the end of gynecologic laparoscopic surgery and prior to trocar removal, 40 mL of Bupivacaine 0.25% is instilled intraperitoneal under direct vision to evaluate its analgesic effect.
  Arms: Intraperitoneal Local Anesthetic Injection (Group B)
Drug: Bupivacaine 0.25% — Before trocar insertion in gynecologic laparoscopic surgery, 5 mL of Bupivacaine 0.25% is infiltrated subcutaneously at each trocar port site to assess its effect on postoperative pain.
  Arms: Port Site Local Anesthetic Injection (Group A)

SUMMARY:
This is a randomized, double-blind, controlled clinical trial evaluating the efficacy of local anesthetic (LA) in reducing postoperative pain in patients undergoing gynecologic laparoscopic surgery. Ninety participants will be randomly assigned into three equal groups: Group A will receive LA injection at the port site, Group B will receive intraperitoneal LA injection, and Group C will serve as the control group with no LA intervention. Postoperative pain will be assessed and compared among the three groups.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged 18 to 60 years

Scheduled for elective gynecological laparoscopic procedures, including:

Evaluation for primary or secondary infertility

Assessment of suspected uterine pathology

Evaluation of Müllerian anomalies

Assessment of suspected tubal or peritoneal pathology requiring diagnostic exploration.

Exclusion Criteria:

Known allergy or hypersensitivity to local anesthetics (e.g., lidocaine or bupivacaine)

Body Mass Index (BMI) ≥ 35 kg/m²

Severe hepatic or renal impairment

Chronic pain conditions requiring regular opioid use

History of major abdominal surgery

Refusal to provide informed consent or to enroll in the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain score assessed using the Visual Analog Scale . | 24 hours after surgery
  Postoperative pain will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.
Time to First Analgesic Request | 24 hours after surgery

SECONDARY OUTCOMES:
Total Analgesic Consumption | within 24 hours after surgery
Patient Satisfaction Score | 24 hours postoperatively
  Patient satisfaction will be measured using a10- point Likert Scale, where 1 = Very Dissatisfied and 10 = Very Satisfied. Higher scores indicate greater satisfaction.
Length of Hospital Stay | From end of surgery until hospital discharge assessed up to 7 days
  The duration (in hours) from the end of surgery to the time of hospital discharge will be recorded. This outcome measures the efficiency of recovery and readiness for discharge.
Time to First Patient Ambulation | Within 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 Months after publication of study results for a year.
Access Criteria: Data will be shared upon reasonable request by contacting the corresponding author. Researchers must sign a data use agreement to access the data.

REFERENCES:
- [Derived] Elsaeed UA, Algyoushy EAFIH, Hatem DLM. Effect of port-site and intraperitoneal local anesthetic injection versus placebo on postoperative pain and recovery after gynecologic laparoscopic surgery: a randomized controlled trial. Sci Rep. 2025 Sep 12;15(1):32466. doi: 10.1038/s41598-025-18389-w. PMID 40940430